CLINICAL TRIAL: NCT05634057
Title: Evaluation of the Efficacy of Anisodamine Hydrobromide Combined With Low-molecular-weight Heparin in the Treatment of Patients With Sepsis
Brief Title: Efficacy of Anisodamine Hydrobromide Combined With Low-molecular-weight Heparin in the Treatment of Patients With Sepsis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chen Ying (Other)
Responsible Party: Sponsor-Investigator, Chen Ying, Research assistant；Junior technician, Beijing Chao Yang Hospital
Organization: Beijing Chao Yang Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Z211100002921061
Record Dates: First submitted 2022-11-09; First posted 2022-12-01 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis | interventions — Heparin

STUDY DESIGN:
Intervention Model Description: The SEPSIS patients will be randomly assigned to four groups in a ratio of 1:1. The groups will consist of the conventional treatment group and the anisodamine hydrobromide combined with heparin treatment group.
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Anisodamine hydrobromide combined with heparin (Experimental): Anisodamine hydrobromide injection + low molecular weight heparin + basic treatment: The dosage of scopolamine butylbromide is 2.0mg/(kg*d), administered via a micro-pump at a constant rate, continuously for 3 days. The dosage range for low molecular weight heparin is limited to 3000-6000U, administered subcutaneously once daily, continuously for 3 days.
  Interventions: Drug: Anisodamine hydrobromide combined with heparin
- conventional therapy (No Intervention): Conventional treatment includes shock treatment, eliminating the cause of the condition, actively treating the primary disease, replenishing blood volume, correcting acid-base imbalances, using vasoactive drugs to maintain blood pressure, and advanced life support as needed, such as the use of a ventilator and bedside blood filtration for organ support.

INTERVENTIONS:
Drug: Anisodamine hydrobromide combined with heparin — The anisodamine hydrobromide combined with heparin treatment group is on the basis of conventional treatment.
  Arms: Anisodamine hydrobromide combined with heparin

SUMMARY:
The study aimed to investigate the effectiveness of anisodamine hydrobromide combined with heparin in the treatment of patients with critical infection, in the hope that the therapy will provide alternatives to the treatment of patients with critical infection.

DETAILED DESCRIPTION:
Objective: The study aimed to investigate the effectiveness of anisodamine hydrobromide combined with heparin in the treatment of patients with critical infection, in the hope that the therapy will provide alternatives to the treatment of patients with critical infection.

Methods: The study is a multi-center randomized controlled clinical trial. Study population will include critically infected patients requiring vasopressor use. The critically infected patients will be randomly assigned to four groups in a ratio of 1:1. The groups will consist of the conventional treatment group and the anisodamine hydrobromide combined with heparin treatment group.

Interim analysis will be performed. The primary study end point is 28-day mortality, and other secondary study endpoint is lactate clearance rate. The investigators will appropriately use chi-square test, student t test or rank sum test to compare the differences between the experimental groups and the control group.

Discussion: The treatment of anisodamine hydrobromide combined with heparin will be better than the conventional treatment. The study will provide new insight into the treatment of patients with critical infection and can help to reduce mortality rate of critically infected patients.

ELIGIBILITY:
Inclusion criteria:

1. Age greater than 18 years;
2. Meets the diagnostic criteria for sepsis according to the "Sepsis-3" ;
3. Patient or their legal representative consents to treatment and signs an informed consent form.

Exclusion criteria:

1. Patients expected to die within 24 hours after enrollment;
2. Contraindications to low molecular weight heparin and scopolamine butylbromide drugs;
3. Patients with thrombotic diseases requiring treatment with low molecular weight heparin;
4. Patients with terminal-stage malignancies, severe immunodeficiency, immunosuppression, severe liver or kidney dysfunction (defined as liver or kidney SOFA score ≥ 3 points), etc.;
5. Pregnant and lactating women;
6. Patients participating in other clinical trials.

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 782 (Estimated)
Dates: Start 2024-01-25 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
28-day mortality | Every patients' survival time will be observed on day 28 after admission.
  The patients will be followed up for 28 days, as our usual hospital length of stay for critically infected patients is 28 days. The investigators will recorded the specific time of death.

SECONDARY OUTCOMES:
Lactate clearance rate | The lactate clearance rate was observed at 6 hours, 24 hours, and 72 hours after admission.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Chaoyang Hospital, Capital Medical University, Beijing, China, China

IPD SHARING:
Plan to Share IPD: No